CLINICAL TRIAL: NCT01691664
Title: Adoptive Cellular Therapy and Radiation Therapy After Surgery in Treating Patients With Esophageal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jun Ren MD, PhD, Director, Capital Medical University Cancer Center, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JR-02
Record Dates: First submitted 2012-09-18; First posted 2012-09-25 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Esophageal Cancer
Keywords: Esophageal Cancer; DC-CIK; immunotherapy; cellular therapy; radiation therapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Only radiation therapy (Active Comparator): Radiotherapy:Patients will be conducted CT simulation, and three-dimensional conformal radiation therapy (3DCRT) or Intensity-modulated radiation therapy(IMRT)was performed. 1.8-2.0 Gy/fraction, 5 fractions a week, with a total dose of 50Gy will be delivered for all patients by 6-MV-X-ray of linear accelerator.
  Interventions: Radiation: Only radiation therapy
- Radiation therapy plus DC-CIK cellular therapy (Experimental): Radiotherapy:Patients will be conducted CT simulation, and three-dimensional conformal radiation therapy (3DCRT) or Intensity-modulated radiation therapy(IMRT)was performed. 1.8-2.0 Gy/fraction, 5 fractions a week, with a total dose of 50Gy will be delivered for all patients by 6-MV-X-ray of linear accelerator.
  DC-CIK cellular therapy:Mononuclear cells were collected aseptically with blood cell separator composition apheresis 3 days before radiation, and cultured DC-CIK cells for 10 days. Cells were infused back to the patients in 3 times between the radiation intermittent period.
  Interventions: Other: Radiation therapy plus DC-CIK cellular therapy

INTERVENTIONS:
Radiation: Only radiation therapy — Patients only radiation therapy after surgery
  Arms: Only radiation therapy
Other: Radiation therapy plus DC-CIK cellular therapy — Patients receive radiation therapy plus DC-CIK cellular therapy after surgery
  Arms: Radiation therapy plus DC-CIK cellular therapy

SUMMARY:
Cytokine-induced killer (CIK) cells show cytolytic activity against tumor. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining Radiation therapy with adoptive cellular therapy after surgery may be more effective than uses radiation therapy alone in treating esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* cytologically or histologically confirmed esophageal carcinoma
* Tumor extension beyond muscularis propria and/or nodal involvement without evidence of M1 disease
* Prior en bloc resection, with curative intent, of all known tumor
* No metastatic disease
* Age: > 18
* Karnofsky performance status ≥ 70
* At least 3 weeks since prior surgery
* Normal functions of heart, lung, liver, kidney and bone marrow
* Blood exams qualified for chemotherapy, which included hemoglobulin ≥9 g/dl, neutrophil ≥1.5×109/L and platelet (PLT) ≥100×109/L, creatinine ≤1.5 UNL
* All patients must be evaluated by a radiation oncologist prior to enrollment to ensure patient is appropriate for radiotherapy
* Informed consent signed

Exclusion Criteria:

* Patients with metastatic disease.
* Patients who are pregnant or nursing.
* Patients with poor bone marrow, liver and kidney functions, which would make radiation therapy intolerable
* Patients with contraindication for irradiation: complete obstruction of esophagus, deep esophageal ulcer, fistula to mediastinum, or haematemesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-09; Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 4 years

SECONDARY OUTCOMES:
quality of life | Initial assessment → months 1,3,6 and 12

OTHER OUTCOMES:
Immunological assessment | Initial assessment, months 1,3,6and 12

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ren, MD, PhD, Principal Investigator — Capital Medical University Cancer Center
Locations (1):
- Beijing Shijitan Hospital, Beijing, Beijing Municipality, China